CLINICAL TRIAL: NCT07049133
Title: Identification Of Toxicity Markers to Trastuzumab-Deruxtecan (T-DXd) In Patients With Advanced Breast Cancer. Tox-DXd: a Prospective, Observational Study
Brief Title: Toxicity Markers to Trastuzumab-Deruxtecan (T-DXd) In Patients With Advanced Breast Cancer
Acronym: Tox-DXd
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: UID 4972; L2-335 (Other: Comitato Etico Territoriale Lombardia 2)
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Trastuzumab-Deruxtecan; ILD/pulmonitis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HER2-positive or HER2- low/ultralow metastatic patient: Candidate to receive T-DXd as per standard practice for HER2-positive or HER2- low/ultralow advanced breast cancer.
  Interventions: Other: T-DXd toxicity marker identification

INTERVENTIONS:
Other: T-DXd toxicity marker identification — to find potential predictive markers associated with T-DXd-related toxicities

SUMMARY:
the anti-Human Epidermal Growth Factor Receptor 2 (HER2) Trastuzumab-Deruxtecan (T-DXd) has shown impressive clinical activity in pretreated patients with metastatic breast cancer (MBC) but is also associated with a non-negligible rate of adverse events that may lead to treatment discontinuation and/or the onset of pneumonitis/interstitial lung disease (ILD)

The aim of the study is to identify and describe potentially predictive markers related to the onset of relevant T-DXd-related toxicities

DETAILED DESCRIPTION:
Despite advanced in diagnosis and in the treatment management, advanced breast cancer (ABC) is still an incurable disease.

Recent pharmaceutical developments have changed treatment algorithms in MBC and have further improved the overall prognosis of patients which exploit the tumor-targeting activity of monoclonal antibodies to deliver at the tumor site potent chemotherapeutic agents that would otherwise be exceedingly toxic if delivered systemically.

Among them, new effective anticancer drugs, such as Trastuzumab-Deruxtecan (T-DXd), have revolutionized the clinical management of HER2-positive and HER2-low ABC. However, this drug is associated with a non-negligible rate of adverse events that can lead to treatment discontinuation and/or the onset of pneumonitis/interstitial lung disease (ILD), a potentially fatal adverse event.

The aim of the study is to identify and describe potentially predictive markers related to the onset of relevant T-DXd-related toxicities (both any grade ILD/pneumonitis and any toxicity of grade ≥3) in a population of patients treated with T-DXd according to standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged at least 18 years.
* Histologically documented invasive breast cancer, either HER2-positive or HER2-low/ultralow.
* Candidate to receive T-DXd as per standard practice.
* Consent for the provision of blood samples for exploratory analyses.

Exclusion Criteria:

* Operable, non-metastatic breast cancer
* Unwillingness to provide additional blood draws

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male or female advanced breast cancer patient, either HER2-positive or HER2-low/ultralow, candidate to receive T-DXd as per standard practice
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of mean levels of cytokine and T-DXd toxicity | 2 years
  cytokine quantification in blood sample collected at baseline and before cycle 3 day 1

SECONDARY OUTCOMES:
Incidence of T-DXd Treatment Adverse Events | 2 years
  Adverse event (AE) collection with particular focus on ILD/pneumonitis and any other Grade 3 (G3) AE
T-DXd activity evaluation | 8 months
  collection of tumor assessment data during T-DXd therapy

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Munzone, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncolgy, Milan, Italy